CLINICAL TRIAL: NCT07222670
Title: A Randomized, Double-Blind, Two-Part, Placebo-Controlled, Multicenter, Phase 2a Study to Evaluate Safety, Tolerability, and Efficacy of INNA-051 as Prophylaxis for Respiratory Tract Illness in Healthy Adults 18 to 45 Years of Age Who Are at Risk for Viral Respiratory Infections
Brief Title: A Study Assessing Safety, Tolerability, and Efficacy of INNA-051 in Preventing Respiratory Illness Due to Viral Infections in Healthy Adults 18 to 45 Years of Age
Acronym: POSITS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ENA Respiratory Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: INNA-051-POC-001
Record Dates: First submitted 2025-10-28; First posted 2025-10-30 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Viral Respiratory Infection; Viral Respiratory Illnesses
Keywords: Respiratory virus; Viral respiratory infection; Viral respiratory illness; Prophylaxis; Intranasal; Viral respiratory disease
MeSH Terms: interventions — INNA-051

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- INNA-051 (Experimental)
  Interventions: Drug: INNA-051
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: INNA-051 — powder nasal spray.
  Arms: INNA-051
Other: Placebo — powder nasal spray.
  Arms: Placebo

SUMMARY:
Acute upper and lower respiratory infections are a major public health problem and a leading cause of morbidity and mortality worldwide. The purpose of this trial is to assess the safety of the investigational agent INNA-051, given intranasally, and its potential effectiveness in reducing the occurrence, severity, and/or the duration of illness resulting from respiratory virus infections. The trial will enroll generally healthy adults (age 18 - 45 years) who are at risk for exposure to viral respiratory infection, for example, due to living conditions or occupation. Participants will be treated with INNA-051 or placebo once weekly for 4 weeks (Part A) or 12 weeks (Part B) during the respiratory virus season.

DETAILED DESCRIPTION:
Viral respiratory infections are associated with significant morbidity and mortality. The diversity of viruses, along with their propensity for mutation, ignited an interest in host-directed therapies that are effective across a wide range of viral pathogens. Toll-like receptors (TLRs) are potential targets for the development of such agents given their central role in host immune defenses.

INNA-051, a TLR2/6 agonist, is being developed as an intranasal innate immune-boosting prophylactic approach for individuals at risk for symptoms and/or complications resulting from respiratory viral infections due to age, occupation, and/or co-morbidities.

This randomized, double-blind, two-part, placebo-controlled, multicenter, Phase 2a trial is designed to evaluate the safety, tolerability, and efficacy of INNA-051 in generally healthy adult participants (age 18 to 45 years, inclusive) who are at increased risk for exposure to viral respiratory infections.

The primary purpose of Part A of the trial is to assess the safety and tolerability of INNA-051 (bilateral intranasal dry powder) in an outpatient setting compared with placebo. In part A of the trial, INNA-051 will be self-administered once weekly for 4 weeks in an outpatient setting during the respiratory virus season.

The purpose of Part B of the trial is to measure the safety, tolerability, and efficacy of INNA-051 bilateral intranasal dry powder compared with placebo in the prevention of symptomatic clinical illness due to RT-qPCR-confirmed viral respiratory infections. In part B of the trial, INNA-051 will be self-administered once weekly for 12 weeks during the North American respiratory virus season.

ELIGIBILITY:
Inclusion Criteria:

* In good general health and without clinically significant medical, psychiatric, chronic or intermittent health conditions.
* At risk for exposure to viral respiratory infection, for example, living in crowded housing, university housing, or military barracks, working in a childcare center or caring for a child aged 10 or less, healthcare workers, factory workers, taxi and bus drivers, grocery clerks, and educators or counselors who work in crowded environments or with multiple exposures with different people daily.
* Agree to use highly effective birth control.

Exclusion Criteria:

* Presence of Type I or Type II diabetes, asthma or other chronic respiratory condition.
* Active infections including Hepatitis B Virus, Hepatitis C Virus, or Human Immunodeficiency (HIV).
* Concurrent participation in another clinical trial involving investigational product or prior receipt of investigational product within 90 days or 5 half-lives of the product.
* Active clinical signs or symptoms of acute respiratory illness (runny nose, sore throat, fever, etc.).
* Received a vaccine against Respiratory Syncytial Virus (RSV) or COVID-19 within 180 days.
* Pregnant or lactating women.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1100 (Estimated)
Dates: Start 2025-12-04 (Actual); Primary Completion 2027-02-09 (Estimated); Study Completion 2027-02-09 (Estimated)

PRIMARY OUTCOMES:
Part A - Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Up to 8 weeks
Part A - Percentage of Participants with TEAEs | Up to 8 weeks
Part A - Number of participants with Serious Adverse Events (SAEs) | Up to 8 weeks
Part A - Percentage of Participants with SAEs | Up to 8 weeks
Part A - Number of Participants with Nasal Irritancy Questionnaire Symptoms (iTNSS Questionnaire) | Up to 4 weeks
Part A - Percentage of Participants with Nasal Irritancy Questionnaire Symptoms (iTNSS Questionnaire) | Up to 4 weeks
Part A - Change in White Blood Cell Count from Baseline | Baseline up to 4 weeks
Part A - Change in Platelet Count from Baseline | Baseline up to 4 weeks
Part A - Change in Hemoglobin from Baseline | Baseline up to 4 weeks
Part A - Change in Alanine Transaminase (ALT) from Baseline | Baseline up to 4 weeks
Part A - Change in Bilirubin (Total) from Baseline | Baseline up to 4 weeks
Part A - Change in Bilirubin (Direct) from Baseline | Baseline up to 4 weeks
Part A - Change in Alkaline Phosphatase (ALP) from Baseline | Baseline up to 4 weeks
Part A - Change in Creatinine from Baseline | Baseline up to 4 weeks
Part A - Change in High Sensitivity C-reactive Protein from Baseline | Baseline up to 4 weeks
Part B - Number of Participants with TEAEs | Up to 16 weeks
Part B - Percentage of Participants with TEAEs | Up to 16 weeks
Part B - Number of Participants with SAEs | Up to 16 weeks
Part B - Percentage of Participants with SAEs | Up to 16 weeks
Part B - Number of Participants with Nasal Irritancy Questionnaire Symptoms (iTNSS Questionnaire) | Up to 12 weeks
Part B - Percentage of Participants with Nasal Irritancy Questionnaire Symptoms (iTNSS Questionnaire) | Up to 12 weeks
Part B - Change in White Blood Cell Count from Baseline | Baseline up to 12 weeks
Part B - Change in Platelet Count from Baseline | Baseline up to 12 weeks
Part B - Change in Hemoglobin from Baseline | Baseline up to 12 weeks
Part B - Change in ALT from Baseline | Baseline up to 12 weeks
Part B - Change in Bilirubin (Total) from Baseline | Baseline up to 12 weeks
Part B - Change in Bilirubin (Direct) from Baseline | Baseline up to 12 weeks
Part B - Change in ALP from Baseline | Baseline up to 12 weeks
Part B - Change in Creatinine from Baseline | Baseline up to 12 weeks
Part B - Change in High Sensitivity C-reactive Protein from Baseline | Baseline up to 12 weeks
Part B - Number of Participants with Reverse Transcription Quantitative Polymerase Chain Reaction (RT-qPCR)-confirmed Symptomatic Viral Respiratory Infections | Up to 12 weeks
Part B - Area Under the Curve (AUC) of the Total Respiratory and Systemic Symptom Scores for Participants with RT-qPCR-confirmed Symptomatic Viral Respiratory Infections | Up to 12 weeks
  The AUC of the total respiratory and systemic symptom scores will be assessed using the respiratory infection intensity and impact questionnaire (RiiQ) for participants with RT-qPCR-confirmed symptomatic viral respiratory infections.

SECONDARY OUTCOMES:
Part B - Number of Participants With RT-qPCR-confirmed Symptomatic Viral Respiratory Infections by Pathogen | Up to 12 weeks
Part B - AUC of the Total Respiratory and Systemic Symptom Scores for Participants with RT-qPCR-confirmed Symptomatic Viral Respiratory Infections by Pathogen | Up to 12 weeks
  The AUC of the total respiratory and systemic symptom scores will be assessed using the RiiQ for participants with RT-qPCR-confirmed symptomatic viral respiratory infections.
Part B - Time to Symptom Resolution in Participants with RT-qPCR-confirmed Symptomatic Viral Respiratory Infections | Up to 12 weeks
  Time to symptom resolution in participants with RT-qPCR-confirmed symptomatic viral respiratory infections will be measured using the RiiQ.
Part B - Duration of Infection for Participants with RT-qPCR-confirmed Symptomatic Viral Respiratory Infections | Up to 12 weeks
  Duration of Infection for participants with RT-qPCR-confirmed symptomatic viral respiratory infections as assessed by time to undetectable viral load measured by RT-qPCR.
Part B - Activities of Daily Living in Participants who have RT-qPCR-Confirmed Symptomatic Viral Respiratory Infections (assessed by EuroQol 5-Dimensions 5-Levels questionnaire [EQ-5D-5L]) | Up to 12 weeks

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Center for Vaccine Development and Global Health (CVD), Baltimore, Maryland
  - Naval Medical Research Command (NMRC), Bethesda, Maryland
  - Accellacare of Raleigh, Raleigh, North Carolina
  - Accellacare of Piedmont HealthCare, Statesville, North Carolina
  - Accellacare - Wilmington, Wilmington, North Carolina

IPD SHARING:
Plan to Share IPD: No